CLINICAL TRIAL: NCT00021268
Title: Phase I Study Of Tocladesine In Patients With Colorectal Carcinoma Following Therapy With 5-FU And Irinotecan
Brief Title: Tocladesine in Treating Patients With Recurrent or Progressive Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: ICN-2000-1; UCLA-0006008; CDR0000068764 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1979
Record Dates: First submitted 2001-07-11; First posted 2003-09-10 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2002-10

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — 8-chloro-cyclic adenosine monophosphate

INTERVENTIONS:
Drug: tocladesine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of tocladesine in treating patients who have recurrent or progressive metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of tocladesine in patients with recurrent or progressive metastatic colorectal cancer.
* Determine the qualitative and quantitative toxicity of this drug in these patients.
* Assess any therapeutic activity in patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive tocladesine IV continuously on days 1-5 and 8-12. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tocladesine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 14 additional patients are treated at this dose level.

PROJECTED ACCRUAL: A total of 3-38 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic carcinoma of the colon or rectum

  * Recurrent or progressive after failing prior fluorouracil and irinotecan chemotherapy, sequentially or in combination, unless unable to tolerate irinotecan
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 5 times ULN
* PT/aPTT no greater than 1.2 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 50 mL/min
* No impaired renal function

Cardiovascular:

* No impaired cardiac function

Other:

* No active infection
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent anticancer drugs
* No concurrent chronic non-steroidal anti-inflammatory agents
* No concurrent chronic therapeutic anticoagulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Rosen, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States